CLINICAL TRIAL: NCT01166308
Title: Randomised Phase I/II Study to Evaluate Carbon Ion Radiotherapy Versus Fractionated Stereotactic Radiotherapy in Patients With Recurrent or Progressive Gliomas: The CINDERELLA Trial
Brief Title: Carbon Ion Radiotherapy for Recurrent Gliomas
Acronym: CINDERELLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINDERELLA; 2009-017352-26 (EudraCT Number)
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Glioma
Keywords: Recurrent Glioma
MeSH Terms: conditions — Glioma | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbon Ion Radiotherapy (Experimental): Carbon Ion Radiotherapy in the RD determined within the Phase I Part of the Trial
  Interventions: Radiation: Carbon Ion Radiotherapy
- Standard Treatment: Fractionated Stereotacitc Radiotherapy (Active Comparator): Standard Precision Radiotherapy performed as Fractionated Stereotactic Radiotherapy (FSRT) up to 36 Gy in single dosis of 2 Gy
  Interventions: Radiation: Fractionated Stereotactic Radiotherapy (FSRT)

INTERVENTIONS:
Radiation: Carbon Ion Radiotherapy — Carbon Ion Radiotherapy in the RD determined within the Phase I part of the Study (10 x 3Gy E to 16 x 3 Gy E)
  Arms: Carbon Ion Radiotherapy
Radiation: Fractionated Stereotactic Radiotherapy (FSRT) — Standard Treatment as Re-Irradiation performed as Fractionated Stereotactic Radiotherapy (FSRT)up to 36 Gy in single doses of 2 Gy
  Arms: Standard Treatment: Fractionated Stereotacitc Radiotherapy

SUMMARY:
Treatment of patients with recurrent glioma includes neurosurgical resection, chemotherapy, or radiation therapy. In most cases, a full course of radiotherapy has been applied after primary diagnosis, therefore application of re-irradiation has to be applied cautiously. With modern precision photon techniques such as fractionated stereotactic radiotherapy (FSRT), a second course of radiotherapy is safe and effective and leads to survival times of 22, 16 and 8 months for recurrent WHO grade II, III and IV tumors.

Carbon ions offer physical and biological characteristics. Due to their inverted dose profile and the high local dose deposition within the Bragg peak precise dose application and sparing of normal tissue is possible. Moreover, in comparison to photons, carbon ions offer an increase relative biological effectiveness (RBE), which can be calculated between 2 and 5 depending on the Glioblastoma (GBM) cell line as well as the endpoint analyzed. Protons, however, offer an RBE which is comparable to photons.

First Japanese Data on the evaluation of carbon ion radiation therapy for the treatment of primary high-grade gliomas showed promising results in a small and heterogeneous patient collective.

In the current Phase I/II-CINDERELLA-trial re-irradiation using carbon ions will be compared to FSRT applied to the area of contrast enhancement representing high-grade tumor areas in patients with recurrent gliomas. Within the Phase I Part of the trial, the Recommended Dose (RD) of carbon ion radiotherapy will be determined in a dose escalation scheme. In the subsequent randomized Phase II part, the RD will be evaluated in the experimental arm, compared to the standard arm, FSRT with a total dose of 36 Gy in single doses of 2 Gy.

Primary endpoint of the Phase I part is toxicity. Primary endpoint of the randomized part II is survival after re-irradiation at 12 months, secondary endpoint is progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* unifocal, supratentorial recurrent glioma
* contrast enhancement on T1-weighted MRI and/or Amino-Acid-PET-positive high-grade tumor areas
* indication re-irradiation
* age ≥ 18 years of age
* Karnofsky Performance Score ≥60
* For women with childbearing potential, (and men) adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* Multifocal Glioma or Gliomatosis cerebri
* refusal of the patients to take part in the study
* previous re-irradiation or prior radiosurgery or prio treatment with interstitial radioactive seeds
* time interval of < 6 months after primary radiotherapy
* Patients who have not yet recovered from acute toxicities of prior therapies
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | at 12 months

SECONDARY OUTCOMES:
Progression-free Survival | at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Department of Radiation Oncology, Heidelberg, Germany

REFERENCES:
- [Derived] Combs SE, Burkholder I, Edler L, Rieken S, Habermehl D, Jakel O, Haberer T, Haselmann R, Unterberg A, Wick W, Debus J. Randomised phase I/II study to evaluate carbon ion radiotherapy versus fractionated stereotactic radiotherapy in patients with recurrent or progressive gliomas: the CINDERELLA trial. BMC Cancer. 2010 Oct 6;10:533. doi: 10.1186/1471-2407-10-533. PMID 20925951